CLINICAL TRIAL: NCT01870778
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase III Study to Evaluate the Efficacy, Safety and Tolerability of Serelaxin When Added to Standard Therapy in Acute Heart Failure Patients
Brief Title: Efficacy, Safety and Tolerability of Serelaxin When Added to Standard Therapy in AHF
Acronym: RELAX-AHF-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRLX030A2301; 2013-001498-25 (EudraCT Number)
Record Dates: First submitted 2013-06-03; First posted 2013-06-06 (Estimated); Results first posted 2018-03-30 (Actual); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Acute Heart Failure
Keywords: acute heart failure,; AHF,; multi-center,; randomized,; double-blind

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Serelaxin (RLX030) (Experimental): Participants received continuous intravenous infusion of serelaxin 30 ug/kg/day for 48 hours.
  Interventions: Drug: RLX030
- Placebo (Placebo Comparator): Participants received continuous intravenous infusion of matching placebo to serelaxin for 48 hours.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RLX030 — 1 mg/mL solution in 6 mL vials
  Arms: Serelaxin (RLX030)
Drug: Placebo — Matching placebo solution to serelaxin
  Arms: Placebo

SUMMARY:
The purpose of the study was to evaluate the efficacy, safety and tolerability of intravenous infusion of serelaxin, when added to standard therapy, in acute heart failure (AHF) patients.

DETAILED DESCRIPTION:
This Phase IIIb outcome study in AHF patients was designed as a multicenter, randomized, double-blind, placebo-controlled, event-driven study in order to assess the efficacy, safety and tolerability of intravenous infusion of serelaxin or placebo. The AHF patients randomized to either serelaxin or placebo in the study were followed for a period of 180 days, and were required to receive standard-of-care background HF management during both the index hospitalization and post discharge according to regional or local guidelines/institutional standards.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female 18 years of age, with body weight ≤160 kg
* Hospitalized for AHF with anticipated requirement of IV therapy for at least 48 hours; AHF is defined as including all of the following measured at any time between presentation (including the emergency department) and the end of screening:

  * Persistent dyspnea at rest or with minimal exertion
  * Pulmonary congestion on chest radiograph
  * B-type natriuretic peptide (BNP) ≥500 pg/mL or N-terminal (NT)-proBNP ≥2000 pg/mL; for patients ≥ 75 years of age or with current atrial fibrillation (at the time of randomization), BNP ≥ 750 pg/mL or NT-proBNP ≥ 3,000 pg/mL
* Systolic BP ≥125 mmHg at the start and at the end of screening
* Able to be randomized within 16 hours from presentation to the hospital, including the emergency department
* Received intravenous furosemide of at least 40 mg total (or equivalent) at any time between presentation (this includes outpatient clinic, ambulance, or hospital including emergency department) and the start of screening for the study for the treatment of the current acute HF episode.

Key Exclusion Criteria:

* Dyspnea primarily due to non-cardiac causes
* Known history of respiratory disorders requiring the daily use of IV or oral steroids (does not include inhaled steroids); need for intubation or the current use of IV or oral steroids for chronic obstructive pulmonary disease (COPD)
* Temperature >38.5°C (oral or equivalent) or sepsis or active infection requiring IV anti-microbial treatment
* Clinical evidence of acute coronary syndrome currently or within 30 days prior to enrollment.
* AHF due to significant arrhythmias, which include any of the following: sustained ventricular tachycardia, bradycardia with sustained ventricular rate <45 beats per minute, or atrial fibrillation/flutter with sustained ventricular response of >130 beats per minute
* Patients with severe renal impairment defined as pre-randomization estimated glomerular filtration rate (eGFR) < 25 mL/min/1.73m2 calculated using the Simplified Modification of Diet in Renal Disease (sMDRD) equation, and/or those receiving current or planned dialysis or ultrafiltration
* Patients with hematocrit <25%, or a history of blood transfusion within the 14 days prior to screening, or active life-threatening GI bleeding.
* Known hepatic impairment (as evidenced by total bilirubin > 3 mg/dL, or increased ammonia levels, if performed) or history of cirrhosis with evidence of portal hypertension such as varices.
* Significant, uncorrected, left ventricular outflow obstruction, such as obstructive hypertrophic cardiomyopathy or severe aortic stenosis (i.e., aortic valve area <1.0 cm2 or mean gradient >40 mmHg on prior or current echocardiogram), and severe mitral stenosis
* Severe aortic insufficiency or severe mitral regurgitation for which surgical or percutaneous intervention is indicated.
* Documented, prior to or at the time of randomization, restrictive amyloid myocardiopathy, OR acute myocarditis or hypertrophic obstructive, restrictive, or constrictive cardiomyopathy (does NOT include restrictive mitral filling patterns seen on Doppler echocardiographic assessments of diastolic function).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6600 (Actual)
Dates: Start 2013-10-02 (Actual); Primary Completion 2017-01-23 (Actual); Study Completion 2017-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (423):
- United States (79):
  - Novartis Investigative Site, Huntsville, Alabama
  - Novartis Investigative Site, Montgomery, Alabama
  - Novartis Investigative Site, Tucson, Arizona
  - Novartis Investigative Site, Anaheim, California
  - Novartis Investigative Site, Fresno, California
  - Novartis Investigative Site, Loma Linda, California
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Northridge, California
  - Novartis Investigative Site, Palo Alto, California
  - Novartis Investigative Site, Sacramento, California
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, Sylmar, California
  - Novartis Investigative Site, Walnut Creek, California
  - Novartis Investigative Site, Colorado Springs, Colorado
  - Novartis Investigative Site, Denver, Colorado
  - Novartis Investigative Site, Hartford, Connecticut
  - Novartis Investigative Site, Atlantis, Florida
  - Novartis Investigative Site, Jacksonville, Florida
  - Novartis Investigative Site, Sanford, Florida
  - Novartis Investigative Site, Sarasota, Florida
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, Winter Haven, Florida
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Marietta, Georgia
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Elk Grove Village, Illinois
  - Novartis Investigative Site, Oakbrook Terrace, Illinois
  - Novartis Investigative Site, Peoria, Illinois
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, Muncie, Indiana
  - Novartis Investigative Site, Kansas City, Kansas
  - Novartis Investigative Site, Alexandria, Louisiana
  - Novartis Investigative Site, Baton Rouge, Louisiana
  - Novartis Investigative Site, Covington, Louisiana
  - Novartis Investigative Site, New Orleans, Louisiana
  - Novartis Investigative Site, Annapolis, Maryland
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Worcester, Massachusetts
  - Novartis Investigative Site, Detroit, Michigan
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, Jackson, Mississippi
  - Novartis Investigative Site, Picayune, Mississippi
  - Novartis Investigative Site, Kansas City, Missouri
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Brooklyn, New York
  - Novartis Investigative Site, Kingston, New York
  - Novartis Investigative Site, New Hyde Park, New York
  - Novartis Investigative Site, Rochester, New York
  - Novartis Investigative Site, Stony Brook, New York
  - Novartis Investigative Site, The Bronx, New York
  - Novartis Investigative Site, Chapel Hill, North Carolina
  - Novartis Investigative Site, Durham, North Carolina
  - Novartis Investigative Site, Raleigh, North Carolina
  - Novartis Investigative Site, Canton, Ohio
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Cleveland, Ohio
  - Novartis Investigative Site, Columbus, Ohio
  - Novartis Investigative Site, Toledo, Ohio
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Abington, Pennsylvania
  - Novartis Investigative Site, Natrona Heights, Pennsylvania
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Wynnewood, Pennsylvania
  - Novartis Investigative Site, Providence, Rhode Island
  - Novartis Investigative Site, Warwick, Rhode Island
  - Novartis Investigative Site, Greenville, South Carolina
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Galveston, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Charlottesville, Virginia
  - Novartis Investigative Site, Falls Church, Virginia
  - Novartis Investigative Site, Lynchburg, Virginia
  - Novartis Investigative Site, Roanoke, Virginia
  - Novartis Investigative Site, Seattle, Washington
  - Novartis Investigative Site, Morgantown, West Virginia
- Argentina (16):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Caba, Buenos Aires
  - Novartis Investigative Site, Carapachay, Buenos Aires
  - Novartis Investigative Site, Coronel Suárez, Buenos Aires
  - Novartis Investigative Site, La Plata, Buenos Aires
  - Novartis Investigative Site, San Martín, Buenos Aires
  - Novartis Investigative Site, San Salvador de Jujuy, Jujuy Province
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, San Miguel de Tucumán, Tucumán Province
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, Corrientes
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, Formosa
  - Novartis Investigative Site, Salta
  - Novartis Investigative Site, San Miguel de Tucumán
  - Novartis Investigative Site, Santa Fe
- Australia (10):
  - Novartis Investigative Site, Camperdown, New South Wales
  - Novartis Investigative Site, Concord, New South Wales
  - Novartis Investigative Site, Randwick, New South Wales
  - Novartis Investigative Site, St Leonards, New South Wales
  - Novartis Investigative Site, Herston, Queensland
  - Novartis Investigative Site, Bedford Park, South Australia
  - Novartis Investigative Site, Geelong, Victoria
  - Novartis Investigative Site, Melbourne, Victoria
  - Novartis Investigative Site, Murdoch, Western Australia
  - Novartis Investigative Site, Perth, Western Australia
- Austria (8):
  - Novartis Investigative Site, Innsbruck, Tyrol
  - Novartis Investigative Site, Braunau am Inn
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Salzburg
  - Novartis Investigative Site, Vienna
  - Novartis Investigative Site, Villach
  - Novartis Investigative Site, Wels
- Belgium (7):
  - Novartis Investigative Site, Aalst
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Genk
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Kortrijk
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Mons
- Brazil (7):
  - Novartis Investigative Site, Goiânia, Goiás
  - Novartis Investigative Site, Curitiba, Paraná
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Ribeirão Preto, São Paulo
  - Novartis Investigative Site, São José do Rio Preto, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
- Bulgaria (6):
  - Novartis Investigative Site, Smolyan, Bulgaria
  - Novartis Investigative Site, Pazardzhik
  - Novartis Investigative Site, Pleven
  - Novartis Investigative Site, Plovdiv
  - Novartis Investigative Site, Sofia
  - Novartis Investigative Site, Varna
- Canada (5):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Sainte-Foy, Quebec
  - Novartis Investigative Site, Thetford-Mines, Quebec
- Chile (2):
  - Novartis Investigative Site, Las Condes, Santiago Metropolitan
  - Novartis Investigative Site, Santiago
- Colombia (3):
  - Novartis Investigative Site, Medellín, Antioquia
  - Novartis Investigative Site, Barranquilla
  - Novartis Investigative Site, Florida Blanca
- Czechia (17):
  - Novartis Investigative Site, Brno-Bohunice, Czech Republic
  - Novartis Investigative Site, Frýdek-Místek, Czech Republic
  - Novartis Investigative Site, Kladno, Czech Republic
  - Novartis Investigative Site, Liberec, Czech Republic
  - Novartis Investigative Site, Pardubice, Czech Republic
  - Novartis Investigative Site, Prague, Czech Republic
  - Novartis Investigative Site, Slaný, Czech Republic
  - Novartis Investigative Site, Ústí nad Labem, Czech Republic
  - Novartis Investigative Site, Ústí nad Orlicí, Czech Republic
  - Novartis Investigative Site, Zlín, Czech Republic
  - Novartis Investigative Site, Hradec Králové, CZE
  - Novartis Investigative Site, Benešov
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Jihlava
  - Novartis Investigative Site, Kolín
  - Novartis Investigative Site, Pilsen
  - Novartis Investigative Site, Prague
- Denmark (3):
  - Novartis Investigative Site, Copenhagen NV
  - Novartis Investigative Site, Glostrup Municipality
  - Novartis Investigative Site, Randers
- France (17):
  - Novartis Investigative Site, Amiens
  - Novartis Investigative Site, Besançon
  - Novartis Investigative Site, Béziers
  - Novartis Investigative Site, Bobigny
  - Novartis Investigative Site, Caen
  - Novartis Investigative Site, Chambray-lès-Tours
  - Novartis Investigative Site, La Tronche
  - Novartis Investigative Site, Le Chesnay
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Nancy
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pessac
  - Novartis Investigative Site, Pontoise
  - Novartis Investigative Site, Rouen
  - Novartis Investigative Site, Saint Herblain - Nantes
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Tourcoing
- Germany (50):
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Bad Krozingen
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bitburg
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Brandenburg
  - Novartis Investigative Site, Bremen
  - Novartis Investigative Site, Coburg
  - Novartis Investigative Site, Detmold
  - Novartis Investigative Site, Dortmund
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Erfurt
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Friedberg
  - Novartis Investigative Site, Füssen
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Greifswald
  - Novartis Investigative Site, Halle
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Heilbronn
  - Novartis Investigative Site, Jena
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Kleve
  - Novartis Investigative Site, Koeln-Nippes
  - Novartis Investigative Site, Langen
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Leverkusen
  - Novartis Investigative Site, Limburg
  - Novartis Investigative Site, Ludwigshafen
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Merseburg
  - Novartis Investigative Site, Mönchengladbach
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Neuwied
  - Novartis Investigative Site, Oldenburg
  - Novartis Investigative Site, Regensburg
  - Novartis Investigative Site, Rüsselsheim am Main
  - Novartis Investigative Site, Tübingen
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Villingen-Schwenningen
  - Novartis Investigative Site, Weiden
  - Novartis Investigative Site, Witten
  - Novartis Investigative Site, Wuppertal
  - Novartis Investigative Site, Würzburg
  - Novartis Investigative Site, Zwickau
- Greece (5):
  - Novartis Investigative Site, Athens, GR
  - Novartis Investigative Site, Larissa, GR
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Chaïdári
  - Novartis Investigative Site, Thessaloniki
- Hungary (10):
  - Novartis Investigative Site, Balatonfüred
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Cegléd
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Kaposvár
  - Novartis Investigative Site, Mátészalka
  - Novartis Investigative Site, Pécs
  - Novartis Investigative Site, Székesfehérvár
  - Novartis Investigative Site, Szombathely
  - Novartis Investigative Site, Zalaegerszeg
- Ireland (2):
  - Novartis Investigative Site, Dublin
  - Novartis Investigative Site, Galway
- Israel (11):
  - Novartis Investigative Site, Lower Galilee, Israel
  - Novartis Investigative Site, Ashkelon
  - Novartis Investigative Site, Hadera
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Nahariya
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Rehovot
  - Novartis Investigative Site, Sefad
  - Novartis Investigative Site, Tel Aviv
  - Novartis Investigative Site, Tel Giborim, Holon
- Italy (25):
  - Novartis Investigative Site, Cortona, AR
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Gavardo, BS
  - Novartis Investigative Site, Bolzano, BZ
  - Novartis Investigative Site, Cremona, CR
  - Novartis Investigative Site, Cona, FE
  - Novartis Investigative Site, Foggia, FG
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Pozzilli, IS
  - Novartis Investigative Site, Monza, MB
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Vimercate, MI
  - Novartis Investigative Site, Modena, MO
  - Novartis Investigative Site, Perugia, PG
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Parma, PR
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Albano Laziale, RM
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Rimini, RN
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Trieste, TS
  - Novartis Investigative Site, Udine, UD
  - Novartis Investigative Site, Novara
- Mexico (5):
  - Novartis Investigative Site, Guadalajara, Jalisco
  - Novartis Investigative Site, Mexico City, Mexico City
  - Novartis Investigative Site, San Luis Potosí City, San Luis Potosí
  - Novartis Investigative Site, Culiacán, Sinaloa
  - Novartis Investigative Site, San Luis Potosí City
- Netherlands (15):
  - Novartis Investigative Site, Sneek, The Netherlands
  - Novartis Investigative Site, Almelo
  - Novartis Investigative Site, Amersfoort
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Arnhem
  - Novartis Investigative Site, Deventer
  - Novartis Investigative Site, Gorinchem
  - Novartis Investigative Site, Groningen
  - Novartis Investigative Site, Haarlem
  - Novartis Investigative Site, Hardenberg
  - Novartis Investigative Site, Maastricht
  - Novartis Investigative Site, Nijmegen
  - Novartis Investigative Site, Rotterdam
  - Novartis Investigative Site, Venlo
  - Novartis Investigative Site, Zutphen
- Novartis Investigative Site, Stavanger, Norway
- Novartis Investigative Site, Lima Cercado, Lima region, Peru
- Poland (12):
  - Novartis Investigative Site, Krakow, POL
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Grodzisk Mazowiecki
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Kłodzko
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Lódz
  - Novartis Investigative Site, Oława
  - Novartis Investigative Site, Puławy
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Wroclaw
  - Novartis Investigative Site, Włocławek
- Portugal (10):
  - Novartis Investigative Site, Carnaxide - Linda-A-Velha, Lisbon District
  - Novartis Investigative Site, Vila Real, Portuigal
  - Novartis Investigative Site, Amadora
  - Novartis Investigative Site, Coimbra
  - Novartis Investigative Site, Covilha
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Penafiel
  - Novartis Investigative Site, Porto
  - Novartis Investigative Site, Viana do Castelo
  - Novartis Investigative Site, Vila Nova de Gaia
- Novartis Investigative Site, Mayagüez, Puerto Rico
- Romania (11):
  - Novartis Investigative Site, Târgu Mureş, Mureș County
  - Novartis Investigative Site, Tg. Mures, Mureș County
  - Novartis Investigative Site, Arad
  - Novartis Investigative Site, Baia Mare
  - Novartis Investigative Site, Brasov
  - Novartis Investigative Site, Brăila
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Craiova
  - Novartis Investigative Site, Oradea
  - Novartis Investigative Site, Piteşti
  - Novartis Investigative Site, Timișoara
- Russia (15):
  - Novartis Investigative Site, Barnaul
  - Novartis Investigative Site, Ivanovo
  - Novartis Investigative Site, Kemerovo
  - Novartis Investigative Site, Kirov
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Novosibirsk
  - Novartis Investigative Site, S.-Petersburg
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Samara
  - Novartis Investigative Site, Saratov
  - Novartis Investigative Site, Tomsk
  - Novartis Investigative Site, Vladimir
  - Novartis Investigative Site, Voronezh
  - Novartis Investigative Site, Yaroslavl
  - Novartis Investigative Site, Yekaterinburg
- Slovakia (12):
  - Novartis Investigative Site, Košice, Slovak Republic
  - Novartis Investigative Site, Liptovský Mikuláš, Slovak Republic
  - Novartis Investigative Site, Topoľčany, Slovak Republic
  - Novartis Investigative Site, Banská Bystrica
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Lučenec
  - Novartis Investigative Site, Martin
  - Novartis Investigative Site, Nitra
  - Novartis Investigative Site, Nové Zámky
  - Novartis Investigative Site, Prešov
  - Novartis Investigative Site, Rimavská Sobota
  - Novartis Investigative Site, Trnava
- South Africa (5):
  - Novartis Investigative Site, Bloemfontein, Free State
  - Novartis Investigative Site, Durban
  - Novartis Investigative Site, Johannesburg
  - Novartis Investigative Site, Umhlanga
  - Novartis Investigative Site, Western Cape
- Spain (19):
  - Novartis Investigative Site, Córdoba, Andalusia
  - Novartis Investigative Site, Marbella, Andalusia
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Sanlúcar de Barrameda, Andalusia
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Barcelona
  - Novartis Investigative Site, Sant Joan Despí, Barcelona
  - Novartis Investigative Site, Villamartín, Cadiz
  - Novartis Investigative Site, León, Castille and León
  - Novartis Investigative Site, Badalona, Catalonia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, A Coruña, Galicia
  - Novartis Investigative Site, Getafe, Madrid
  - Novartis Investigative Site, Majadahonda, Madrid
  - Novartis Investigative Site, El Palmar, Murcia
  - Novartis Investigative Site, Alicante, Valencia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
- Sweden (5):
  - Novartis Investigative Site, Jönköping
  - Novartis Investigative Site, Linköping
  - Novartis Investigative Site, Mölndal
  - Novartis Investigative Site, Stockholm
  - Novartis Investigative Site, Uppsala
- Switzerland (4):
  - Novartis Investigative Site, Basel
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Lausanne
  - Novartis Investigative Site, Sankt Gallen
- Turkey (Türkiye) (7):
  - Novartis Investigative Site, Pendik / Istanbul, Turkey
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Haydarpasa/Istanbul
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Kocaeli
  - Novartis Investigative Site, Mersin
  - Novartis Investigative Site, Sivas
- United Kingdom (17):
  - Novartis Investigative Site, High Wycombe, Buckinghamshire
  - Novartis Investigative Site, Torquay, Devon
  - Novartis Investigative Site, Basingstoke, Hampshire
  - Novartis Investigative Site, Nottingham, Hampshire
  - Novartis Investigative Site, Blackburn, Lancashire
  - Novartis Investigative Site, Hardwick, Stockton On Tees
  - Novartis Investigative Site, Dudley, West Midlands
  - Novartis Investigative Site, Blackpool
  - Novartis Investigative Site, Edinburgh
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, Kettering
  - Novartis Investigative Site, Leicester
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Portsmouth
  - Novartis Investigative Site, Swindon

REFERENCES:
- [Derived] Ravera A, Qin H, Ter Maaten JM, Santema BT, Adamo M, Ponikowski P, Cotter G, Davison BA, Felker GM, Filippatos GS, Pang PS, Greenberg BH, Gimpelewicz C, Severin T, Teerkink JR, Voors AA, Metra M. Clinical Presentation, Biomarker Trajectories, and Outcomes in Women and Men Hospitalized for Acute Heart Failure. JACC Heart Fail. 2025 Oct;13(10):102524. doi: 10.1016/j.jchf.2025.102524. Epub 2025 Aug 21. PMID 40845614
- [Derived] Pagnesi M, Staal L, Ter Maaten JM, Beldhuis IE, Cotter G, Davison BA, Jongs N, Felker GM, Filippatos G, Greenberg BH, Pang PS, Ponikowski P, Lombardi CM, Adamo M, Severin T, Gimpelewicz C, Voors AA, Teerlink JR, Metra M. Decongestion and Outcomes in Patients Hospitalized for Acute Heart Failure: Insights From the RELAX-AHF-2 Trial. JACC Heart Fail. 2025 Mar;13(3):414-429. doi: 10.1016/j.jchf.2024.09.013. Epub 2024 Nov 27. PMID 39614837
- [Derived] Grand J, Miger K, Sajadieh A, Kober L, Torp-Pedersen C, Ertl G, Lopez-Sendon J, Pietro Maggioni A, Teerlink JR, Sato N, Gimpelewicz C, Metra M, Holbro T, Nielsen OW. Blood Pressure Drops During Hospitalization for Acute Heart Failure Treated With Serelaxin: A Patient-Level Analysis of 4 Randomized Controlled Trials. Circ Heart Fail. 2022 Apr;15(4):e009199. doi: 10.1161/CIRCHEARTFAILURE.121.009199. Epub 2022 Feb 21. PMID 35184572
- [Derived] Matsue Y, Sama IE, Postmus D, Metra M, Greenberg BH, Cotter G, Davison BA, Felker GM, Filippatos G, Pang P, Ponikowski P, Severin T, Gimpelewicz C, Voors AA, Teerlink JR. Association of Early Blood Pressure Decrease and Renal Function With Prognosis in Acute Heart Failure. JACC Heart Fail. 2021 Dec;9(12):890-903. doi: 10.1016/j.jchf.2021.07.001. Epub 2021 Oct 6. PMID 34627724
- [Derived] Grand J, Miger K, Sajadieh A, Kober L, Torp-Pedersen C, Ertl G, Lopez-Sendon J, Pietro Maggioni A, Teerlink JR, Sato N, Gimpelewicz C, Metra M, Holbro T, Nielsen OW. Systolic Blood Pressure and Outcome in Patients Admitted With Acute Heart Failure: An Analysis of Individual Patient Data From 4 Randomized Clinical Trials. J Am Heart Assoc. 2021 Sep 21;10(18):e022288. doi: 10.1161/JAHA.121.022288. Epub 2021 Sep 13. PMID 34514815
- [Derived] Loungani RS, Teerlink JR, Metra M, Allen LA, Butler J, Carson PE, Chen CW, Cotter G, Davison BA, Eapen ZJ, Filippatos GS, Gimpelewicz C, Greenberg B, Holbro T, Januzzi JL Jr, Lanfear DE, Pang PS, Pina IL, Ponikowski P, Miller AB, Voors AA, Felker GM. Cause of Death in Patients With Acute Heart Failure: Insights From RELAX-AHF-2. JACC Heart Fail. 2020 Dec;8(12):999-1008. doi: 10.1016/j.jchf.2020.09.010. Epub 2020 Nov 11. PMID 33189635
- [Derived] Metra M, Teerlink JR, Cotter G, Davison BA, Felker GM, Filippatos G, Greenberg BH, Pang PS, Ponikowski P, Voors AA, Adams KF, Anker SD, Arias-Mendoza A, Avendano P, Bacal F, Bohm M, Bortman G, Cleland JGF, Cohen-Solal A, Crespo-Leiro MG, Dorobantu M, Echeverria LE, Ferrari R, Goland S, Goncalvesova E, Goudev A, Kober L, Lema-Osores J, Levy PD, McDonald K, Manga P, Merkely B, Mueller C, Pieske B, Silva-Cardoso J, Spinar J, Squire I, Stepinska J, Van Mieghem W, von Lewinski D, Wikstrom G, Yilmaz MB, Hagner N, Holbro T, Hua TA, Sabarwal SV, Severin T, Szecsody P, Gimpelewicz C; RELAX-AHF-2 Committees Investigators. Effects of Serelaxin in Patients with Acute Heart Failure. N Engl J Med. 2019 Aug 22;381(8):716-726. doi: 10.1056/NEJMoa1801291. PMID 31433919
- [Derived] Teerlink JR, Voors AA, Ponikowski P, Pang PS, Greenberg BH, Filippatos G, Felker GM, Davison BA, Cotter G, Gimpelewicz C, Boer-Martins L, Wernsing M, Hua TA, Severin T, Metra M. Serelaxin in addition to standard therapy in acute heart failure: rationale and design of the RELAX-AHF-2 study. Eur J Heart Fail. 2017 Jun;19(6):800-809. doi: 10.1002/ejhf.830. Epub 2017 Apr 28. PMID 28452195

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 6600 participants were randomized into the trial. Only 6545 participants were eligible for analysis. Therefore, the participants flow and baseline characteristics are based on 6545 participants.
Period: Overall Study
Arm/Group | Serelaxin (RLX030) | Placebo
Started | 3274 | 3271
Safety Set | 3257 | 3248
Full Analysis Set | 3274 | 3271
Biomarker Analysis Set | 521 | 510
Completed | 3266 | 3262
Not Completed | 8 | 9
Not completed — Withdrawal by Subject | 8 | 7
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Serelaxin (RLX030) | Placebo | Total
Number analyzed (Participants) | 3274 | 3271 | 6545
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.1 (11.24) | 72.8 (11.17) | 73.0 (11.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1296 | 1341 | 2637
  Male | 1978 | 1930 | 3908
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 13 | 18 | 31
  Asian | 14 | 16 | 30
  Native Hawaiian or Other Pacific Islander | 4 | 4 | 8
  Black or African American | 163 | 171 | 334
  White | 3017 | 2999 | 6016
  More than one race | 46 | 46 | 92
  Unknown or Not Reported | 17 | 17 | 34

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Confirmed Cardiovascular (CV) Death Through Day 180
Description: The percentage of participants with an adjudicated CV death through day 180 was assessed.
Time Frame: 180 days
Population: The Full Analysis Set, which included all randomized participants who were not mis-randomized or excluded due to GCP reasons, was analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Serelaxin (RLX030) | Placebo
Number analyzed (Participants) | 3274 | 3271
Percentage of participants | 8.7 | 8.9
Statistical Analysis 1: Comparison: Serelaxin (RLX030) vs Placebo; Test type: Superiority; p = 0.3857, Log Rank — Adjusted alpha p-value based on multiple testing procedure; One-sided p-value; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.83 to 1.15]

2. Primary Outcome: Percentage of Participants With Worsening of Heart Failure (WHF) Through Day 5
Description: The percentage of participants with WHF through day 5 was assessed.
Time Frame: Day 5
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Serelaxin (RLX030) | Placebo
Number analyzed (Participants) | 3274 | 3271
Percentage of participants | 6.9 | 7.7
Statistical Analysis 1: Comparison: Serelaxin (RLX030) vs Placebo; Test type: Superiority; p = 0.0968, Gehan's generalized Wilcoxon test — Adjusted p-value based on multiple testing procedure; One-sided p-value; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.75 to 1.07]

3. Secondary Outcome: Percentage of Participants With All-cause Death Through Day 180
Description: The percentage of participants with all-cause death through day 180 was assessed.
Time Frame: 180 days
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Serelaxin (RLX030) | Placebo
Number analyzed (Participants) | 3274 | 3271
Percentage of participants | 11.2 | 11.9
Statistical Analysis 1: Comparison: Serelaxin (RLX030) vs Placebo; Test type: Superiority; p = 0.3890, Log Rank; 2-sided p-value; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.81 to 1.08]

4. Secondary Outcome: Length of Total Hospital Stay (LOS) During the Index Acute Heart Failure (AHF) Hospitalization
Description: Length of stay was defined as the index hospitalization discharge date and time minus the baseline date and time plus 1 day.
Time Frame: 180 days (Participants still in the hospital at Day 60 were censored at Day 60)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Serelaxin (RLX030) | Placebo
Number analyzed (Participants) | 3274 | 3271
days | 9.362 (9.3581) | 9.545 (9.6739)
Statistical Analysis 1: Comparison: Serelaxin (RLX030) vs Placebo; Test type: Superiority; p = 0.2204, Wilcoxon rank sum test — Based on multiple testing procedure; One-sided p-value

5. Secondary Outcome: Percentage of Participants With First Occurrence of Adjudicated CV Death or Adjudicated Re-hospitalization
Description: The percentage of participants with adjudicated CV death or adjudicated re-hospitalization through day 180 was assessed.
Time Frame: 180 days
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Serelaxin (RLX030) | Placebo
Number analyzed (Participants) | 3274 | 3271
Percentage of participants | 24.3 | 24.9
Statistical Analysis 1: Comparison: Serelaxin (RLX030) vs Placebo; Test type: Superiority; p = 0.2744, Log Rank — Adjusted p-value based on multiple testing procedure; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.88 to 1.07]

6. Secondary Outcome: Length of Intensive Care Unit (ICU) and/or Coronary Care Unit (CCU) Stay for the Index AHF Hospitalization
Description: Length of stay was defined as the hospitalization discharge date and the time minus the baseline date and time plus 1 day.
Time Frame: 180 days (Patients still in the hospital at Day 60 were censored at Day 60)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Serelaxin (RLX030) | Placebo
Number analyzed (Participants) | 3274 | 3271
days | 3.8 (8.29) | 4.1 (8.77)
Statistical Analysis 1: Comparison: Serelaxin (RLX030) vs Placebo; Test type: Superiority; p = 0.2103, Wilcoxon rank sum test; 2-sided p-value

7. Secondary Outcome: Percentage of Participants With First Improvement Since Baseline in Congestive Signs and Symptoms of Heart Failure
Description: The percentage of participants with first improvement since baseline in congestive signs and symptoms was assessed. The signs and symptoms included exertional dyspnea, orthopnea, rales, jugular venous pressure and peripheral edema/pre-sacral edema.
Time Frame: From baseline to Day 5
Population: The Full Analysis Set, which included all randomized participants who were not mis-randomized or excluded due to GCP reasons, was considered for the analysis. For each symptom, only participants with observed baseline signs and symptoms and non-missing baseline and post baseline signs and symptoms were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Serelaxin (RLX030) | Placebo
Number analyzed (Participants) | 3044 | 3039
Percentage of participants
  Exertional dyspnea | 94.1 | 92.6
  Orthopnea: number analyzed (Participants) | 2937 | 2967
  Orthopnea | 92.9 | 91.2
  Rales: number analyzed (Participants) | 2888 | 2877
  Rales | 94.1 | 93.7
  Jugular venous pressure: number analyzed (Participants) | 2054 | 2034
  Jugular venous pressure | 90.4 | 88.0
  Peripheral edema, pre-sacral edema: number analyzed (Participants) | 2597 | 2622
  Peripheral edema, pre-sacral edema | 91.6 | 90.7
Statistical Analysis 1: Comparison: Serelaxin (RLX030) vs Placebo; Exertional dyspnea; Test type: Superiority; p = 0.0050, Log Rank; 2-sided p-value; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [1.02 to 1.14]
Statistical Analysis 2: Comparison: Serelaxin (RLX030) vs Placebo; Orthopnea; Test type: Superiority; p = 0.0051, Log Rank; 2-sided p-value; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [1.02 to 1.14]
Statistical Analysis 3: Comparison: Serelaxin (RLX030) vs Placebo; Rales; Test type: Superiority; p = 0.9962, Log Rank; 2-sided p-value; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.95 to 1.05]
Statistical Analysis 4: Comparison: Serelaxin (RLX030) vs Placebo; Jugular venous pressure; Test type: Superiority; p = 0.0196, Log Rank; 2-sided p-value; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [1.01 to 1.15]
Statistical Analysis 5: Comparison: Serelaxin (RLX030) vs Placebo; Peripheral edema, pre-sacral edema; Test type: Superiority; p = 0.2158, Log Rank; 2-sided p-value; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.98 to 1.10]

8. Secondary Outcome: Change From Baseline in hsTroponin T Biomarker
Description: Blood samples were collected to assess the change from baseline in hsTroponin T. The geometric least square mean (LSM) of the ratio of the post-baseline value to the baseline value is presented.
Time Frame: Baseline, Day 2, Day 5 and Day 14
Population: Participants from the biomarker analysis set, who had both baseline and post baseline values for a given time point, were analyzed at that time point.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ug/L
Arm/Group | Serelaxin (RLX030) | Placebo
Number analyzed (Participants) | 521 | 510
ug/L
  Day 2: number analyzed (Participants) | 464 | 459
  Day 2 | 0.9808 [0.9452 to 1.0177] | 1.0432 [1.0052 to 1.0827]
  Day 5: number analyzed (Participants) | 458 | 449
  Day 5 | 0.9589 [0.9116 to 1.0087] | 1.0678 [1.0148 to 1.1237]
  Day 14: number analyzed (Participants) | 436 | 418
  Day 14 | 0.7813 [0.7374 to 0.8278] | 0.8611 [0.8119 to 0.9132]
Statistical Analysis 1: Comparison: Serelaxin (RLX030) vs Placebo; Day 2; Test type: Superiority; p = 0.0209, Repeated measures model; Ratio of RLX030 to placebo = 0.9401, 95% CI 2-sided [0.8921 to 0.9907]
Statistical Analysis 2: Comparison: Serelaxin (RLX030) vs Placebo; Day 5; Test type: Superiority; p = 0.0034, Repeated measures model; Ratio of RLX030 to placebo = 0.8980, 95% CI 2-sided [0.8358 to 0.9649]
Statistical Analysis 3: Comparison: Serelaxin (RLX030) vs Placebo; Day 14; Test type: Superiority; p = 0.0209, Repeated measures model; Ratio of RLX030 to placebo = 0.9074, 95% CI 2-sided [0.8355 to 0.9854]

9. Secondary Outcome: Change From Baseline in NT-proBNP Biomarker
Description: Blood samples were collected to assess the change from baseline in NT-proBNP. The ratio of the post-baseline value to the baseline value is presented.
Time Frame: Baseline, Day 2, Day 5 and Day 14
Population: as for outcome 8
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Serelaxin (RLX030) | Placebo
Number analyzed (Participants) | 521 | 510
pg/mL
  Day 2: number analyzed (Participants) | 472 | 465
  Day 2 | 0.4902 [0.4609 to 0.5214] | 0.5702 [0.5358 to 0.6068]
  Day 5: number analyzed (Participants) | 465 | 455
  Day 5 | 0.4249 [0.3950 to 0.4570] | 0.4454 [0.4138 to 0.4794]
  Day 14: number analyzed (Participants) | 446 | 429
  Day 14 | 0.4265 [0.3957 to 0.4596] | 0.4469 [0.4143 to 0.4822]
Statistical Analysis 1: Comparison: Serelaxin (RLX030) vs Placebo; Day 2; Test type: Superiority; p = 0.0007, Repeated measures model; Ratio of RLX030 to placebo = 0.8597, 95% CI 2-sided [0.7876 to 0.9385]
Statistical Analysis 2: Comparison: Serelaxin (RLX030) vs Placebo; Day 5; Test type: Superiority; p = 0.3709, Repeated measures model; Ratio of RLX030 to placebo = 0.9539, 95% CI 2-sided [0.8600 to 1.0579]
Statistical Analysis 3: Comparison: Serelaxin (RLX030) vs Placebo; Day 14; Test type: Superiority; p = 0.3893, Repeated measures model; Ratio of RLX030 to placebo = 0.9543, 95% CI 2-sided [0.8578 to 1.0617]

10. Secondary Outcome: Change From Baseline in Cystatin C Biomarker
Description: Blood samples were collected to assess the change from baseline in Cystatin C. The ratio of the post-baseline value to the baseline value is presented.
Time Frame: Baseline, Day 2, Day 5 and Day 14
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/L
Arm/Group | Serelaxin (RLX030) | Placebo
Number analyzed (Participants) | 521 | 510
mg/L
  Day 2: number analyzed (Participants) | 474 | 465
  Day 2 | 1.0261 [1.0119 to 1.0406] | 1.0648 [1.0499 to 1.0799]
  Day 5: number analyzed (Participants) | 467 | 456
  Day 5 | 1.1171 [1.0976 to 1.1369] | 1.1259 [1.1061 to 1.1461]
  Day 14: number analyzed (Participants) | 445 | 432
  Day 14 | 1.1186 [1.0949 to 1.1429] | 1.1342 [1.1098 to 1.1591]
Statistical Analysis 1: Comparison: Serelaxin (RLX030) vs Placebo; Day 2; Test type: Superiority; p = 0.0003, Repeated measures model; Ratio of RLX030 to placebo = 0.9637, 95% CI 2-sided [0.9447 to 0.9830]
Statistical Analysis 2: Comparison: Serelaxin (RLX030) vs Placebo; Day 5; Test type: Superiority; p = 0.5361, Repeated measures model; Ratio of RLX030 to placebo = 0.9922, 95% CI 2-sided [0.9677 to 1.0172]
Statistical Analysis 3: Comparison: Serelaxin (RLX030) vs Placebo; Day 14; Test type: Superiority; p = 0.3750, Repeated measures model; Ratio of RLX030 to placebo = 0.9863, 95% CI 2-sided [0.9567 to 1.0169]

ADVERSE EVENTS:
Time Frame: up to 180 days
Arm/Group | Serelaxin (RLX030) | Placebo
All-Cause Mortality (participants affected / at risk) | 363/3257 | 386/3248
Serious Adverse Events (participants affected / at risk) | 412/3257 | 424/3248
Other Adverse Events (participants affected / at risk) | 1336/3257 | 1277/3248
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Serelaxin (RLX030) (N=3257) | Placebo (N=3248)
Anaemia (Blood and lymphatic system disorders) | 7 | 7
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 1
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 3
Acute left ventricular failure (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 14 | 12
Angina pectoris (Cardiac disorders) | 1 | 7
Angina unstable (Cardiac disorders) | 2 | 2
Aortic valve incompetence (Cardiac disorders) | 1 | 2
Aortic valve stenosis (Cardiac disorders) | 4 | 9
Arrhythmia (Cardiac disorders) | 0 | 2
Arteriosclerosis coronary artery (Cardiac disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 10 | 13
Atrial flutter (Cardiac disorders) | 2 | 2
Atrial thrombosis (Cardiac disorders) | 0 | 1
Atrioventricular block (Cardiac disorders) | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 5 | 2
Atrioventricular block second degree (Cardiac disorders) | 0 | 1
Atrioventricular dissociation (Cardiac disorders) | 1 | 0
Bradyarrhythmia (Cardiac disorders) | 1 | 1
Bradycardia (Cardiac disorders) | 4 | 4
Cardiac arrest (Cardiac disorders) | 4 | 9
Cardiac failure (Cardiac disorders) | 62 | 68
Cardiac failure acute (Cardiac disorders) | 14 | 8
Cardiac failure chronic (Cardiac disorders) | 2 | 3
Cardiac failure congestive (Cardiac disorders) | 12 | 9
Cardio-respiratory arrest (Cardiac disorders) | 2 | 2
Cardiogenic shock (Cardiac disorders) | 5 | 6
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Cardiorenal syndrome (Cardiac disorders) | 1 | 2
Chordae tendinae rupture (Cardiac disorders) | 2 | 1
Congestive cardiomyopathy (Cardiac disorders) | 0 | 2
Coronary artery disease (Cardiac disorders) | 17 | 12
Coronary artery occlusion (Cardiac disorders) | 1 | 1
Coronary artery perforation (Cardiac disorders) | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 5 | 2
Defect conduction intraventricular (Cardiac disorders) | 0 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 2 | 0
Mitral valve incompetence (Cardiac disorders) | 5 | 5
Mitral valve stenosis (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 3 | 4
Myocardial ischaemia (Cardiac disorders) | 2 | 3
Pericarditis (Cardiac disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 2
Sinus node dysfunction (Cardiac disorders) | 1 | 2
Supraventricular tachycardia (Cardiac disorders) | 1 | 2
Tachyarrhythmia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Torsade de pointes (Cardiac disorders) | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 1 | 1
Ventricular fibrillation (Cardiac disorders) | 4 | 6
Ventricular tachycardia (Cardiac disorders) | 14 | 11
Hyperthyroidism (Endocrine disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0
Gastroduodenal ulcer (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 2
Haematochezia (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 2 | 0
Ileus paralytic (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 1
Intestinal stenosis (Gastrointestinal disorders) | 0 | 1
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 1
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Subileus (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Cardiac death (General disorders) | 0 | 2
Drug effect increased (General disorders) | 1 | 0
Extravasation (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 1 | 0
Inflammation (General disorders) | 1 | 0
Infusion site phlebitis (General disorders) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 4 | 1
Non-cardiac chest pain (General disorders) | 2 | 0
Pyrexia (General disorders) | 0 | 1
Sudden cardiac death (General disorders) | 3 | 6
Sudden death (General disorders) | 0 | 1
Vascular stent occlusion (General disorders) | 0 | 1
Alcoholic liver disease (Hepatobiliary disorders) | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1
Hepatic congestion (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 2 | 3
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Hepatocellular injury (Hepatobiliary disorders) | 2 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 1 | 0
Liver injury (Hepatobiliary disorders) | 1 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Abdominal abscess (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Arthritis bacterial (Infections and infestations) | 1 | 0
Aspergilloma (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 9 | 4
Cellulitis (Infections and infestations) | 0 | 1
Cholecystitis infective (Infections and infestations) | 1 | 0
Chronic hepatitis B (Infections and infestations) | 1 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 1
Cystitis (Infections and infestations) | 3 | 1
Cystitis bacterial (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Enterocolitis bacterial (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 2
Gastroenteritis clostridial (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Intervertebral discitis (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 2 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Nosocomial infection (Infections and infestations) | 1 | 0
Orchitis (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0
Pneumococcal sepsis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 34 | 32
Pneumonia streptococcal (Infections and infestations) | 1 | 0
Pulmonary sepsis (Infections and infestations) | 1 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 6 | 8
Septic shock (Infections and infestations) | 4 | 2
Staphylococcal bacteraemia (Infections and infestations) | 2 | 3
Staphylococcal infection (Infections and infestations) | 0 | 1
Streptococcal bacteraemia (Infections and infestations) | 1 | 0
Streptococcal sepsis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 13 | 5
Urinary tract infection pseudomonal (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 1 | 3
Aortic restenosis (Injury, poisoning and procedural complications) | 1 | 0
Cardiac valve replacement complication (Injury, poisoning and procedural complications) | 0 | 1
Coronary artery restenosis (Injury, poisoning and procedural complications) | 2 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2 | 0
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 1 | 0
Procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Procedural hypotension (Injury, poisoning and procedural complications) | 1 | 0
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 2
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 2 | 0
Blood creatinine increased (Investigations) | 1 | 2
Blood pressure decreased (Investigations) | 0 | 2
C-reactive protein increased (Investigations) | 1 | 1
Cardiac output decreased (Investigations) | 1 | 0
Ejection fraction decreased (Investigations) | 2 | 2
Electrocardiogram T wave inversion (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 3 | 1
Liver function test increased (Investigations) | 0 | 1
Oxygen saturation decreased (Investigations) | 1 | 0
Troponin increased (Investigations) | 1 | 1
Vascular resistance pulmonary increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Metabolic alkalosis (Metabolism and nutrition disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Facial asymmetry (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Mediastinum neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Waldenstrom's macroglobulinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Altered state of consciousness (Nervous system disorders) | 1 | 0
Aphasia (Nervous system disorders) | 1 | 1
Brain stem stroke (Nervous system disorders) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Carotid sinus syndrome (Nervous system disorders) | 1 | 1
Cerebral artery embolism (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 2 | 3
Cognitive disorder (Nervous system disorders) | 0 | 1
Dementia (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1
Embolic stroke (Nervous system disorders) | 1 | 1
Epilepsy (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 1
Hypercapnic coma (Nervous system disorders) | 0 | 1
Ischaemic cerebral infarction (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 11 | 16
Loss of consciousness (Nervous system disorders) | 1 | 0
Muscle contractions involuntary (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 2 | 0
Radiculopathy (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 2 | 0
Somnolence (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 5 | 3
Transient ischaemic attack (Nervous system disorders) | 6 | 1
Vascular encephalopathy (Nervous system disorders) | 1 | 0
Device battery issue (Product Issues) | 1 | 0
Device leakage (Product Issues) | 1 | 0
Device malfunction (Product Issues) | 0 | 1
Acute psychosis (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 2 | 1
Delirium (Psychiatric disorders) | 2 | 2
Delirium tremens (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 20 | 25
Anuria (Renal and urinary disorders) | 2 | 0
Azotaemia (Renal and urinary disorders) | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 4 | 3
Haematuria (Renal and urinary disorders) | 1 | 1
Nephropathy toxic (Renal and urinary disorders) | 0 | 6
Nephrotic syndrome (Renal and urinary disorders) | 1 | 1
Oliguria (Renal and urinary disorders) | 1 | 1
Prerenal failure (Renal and urinary disorders) | 1 | 0
Renal artery stenosis (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 10 | 16
Renal impairment (Renal and urinary disorders) | 13 | 9
Renal mass (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Acquired phimosis (Reproductive system and breast disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary cavitation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 7
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 | 10
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Panniculitis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 2
Cardioversion (Surgical and medical procedures) | 1 | 0
Coronary artery bypass (Surgical and medical procedures) | 1 | 0
Toe amputation (Surgical and medical procedures) | 0 | 1
Aortic aneurysm (Vascular disorders) | 0 | 1
Aortic aneurysm rupture (Vascular disorders) | 1 | 0
Aortic dissection (Vascular disorders) | 1 | 0
Arterial stenosis (Vascular disorders) | 0 | 1
Arteriosclerosis (Vascular disorders) | 0 | 2
Arteriovenous fistula (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 3
Hypertensive crisis (Vascular disorders) | 3 | 1
Hypotension (Vascular disorders) | 14 | 9
Hypovolaemic shock (Vascular disorders) | 0 | 1
Iliac artery embolism (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1
Peripheral embolism (Vascular disorders) | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 1
Phlebitis (Vascular disorders) | 0 | 1
Shock (Vascular disorders) | 1 | 0
Subclavian steal syndrome (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Serelaxin (RLX030) (N=3257) | Placebo (N=3248)
Anaemia (Blood and lymphatic system disorders) | 48 | 47
Angina pectoris (Cardiac disorders) | 17 | 15
Aortic valve incompetence (Cardiac disorders) | 21 | 25
Aortic valve stenosis (Cardiac disorders) | 23 | 13
Atrial fibrillation (Cardiac disorders) | 46 | 45
Bradycardia (Cardiac disorders) | 23 | 22
Cardiac failure (Cardiac disorders) | 162 | 185
Mitral valve incompetence (Cardiac disorders) | 52 | 47
Tricuspid valve incompetence (Cardiac disorders) | 30 | 21
Ventricular tachycardia (Cardiac disorders) | 37 | 24
Abdominal pain (Gastrointestinal disorders) | 18 | 19
Constipation (Gastrointestinal disorders) | 70 | 57
Diarrhoea (Gastrointestinal disorders) | 44 | 52
Nausea (Gastrointestinal disorders) | 59 | 51
Vomiting (Gastrointestinal disorders) | 30 | 24
Non-cardiac chest pain (General disorders) | 12 | 20
Pyrexia (General disorders) | 31 | 41
Bronchitis (Infections and infestations) | 30 | 47
Cystitis (Infections and infestations) | 18 | 7
Pneumonia (Infections and infestations) | 17 | 22
Urinary tract infection (Infections and infestations) | 58 | 68
Blood creatinine increased (Investigations) | 36 | 49
Blood potassium decreased (Investigations) | 15 | 20
Blood pressure decreased (Investigations) | 36 | 23
Blood pressure systolic decreased (Investigations) | 29 | 24
Blood urea increased (Investigations) | 24 | 25
Gout (Metabolism and nutrition disorders) | 16 | 28
Hyperglycaemia (Metabolism and nutrition disorders) | 25 | 17
Hyperkalaemia (Metabolism and nutrition disorders) | 40 | 36
Hyperuricaemia (Metabolism and nutrition disorders) | 25 | 21
Hypoglycaemia (Metabolism and nutrition disorders) | 29 | 22
Hypokalaemia (Metabolism and nutrition disorders) | 263 | 241
Hyponatraemia (Metabolism and nutrition disorders) | 19 | 13
Arthralgia (Musculoskeletal and connective tissue disorders) | 25 | 21
Back pain (Musculoskeletal and connective tissue disorders) | 22 | 26
Muscle spasms (Musculoskeletal and connective tissue disorders) | 79 | 49
Pain in extremity (Musculoskeletal and connective tissue disorders) | 27 | 32
Dizziness (Nervous system disorders) | 27 | 17
Headache (Nervous system disorders) | 74 | 92
Anxiety (Psychiatric disorders) | 16 | 30
Confusional state (Psychiatric disorders) | 25 | 28
Insomnia (Psychiatric disorders) | 42 | 48
Acute kidney injury (Renal and urinary disorders) | 35 | 34
Haematuria (Renal and urinary disorders) | 20 | 20
Renal failure (Renal and urinary disorders) | 42 | 46
Renal impairment (Renal and urinary disorders) | 48 | 55
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 6 | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 41 | 36
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 17 | 15
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 19 | 14
Hypertension (Vascular disorders) | 23 | 37
Hypotension (Vascular disorders) | 69 | 58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-03-03): https://cdn.clinicaltrials.gov/large-docs/78/NCT01870778/SAP_000.pdf
  • Study Protocol (2015-02-18): https://cdn.clinicaltrials.gov/large-docs/78/NCT01870778/Prot_001.pdf